CLINICAL TRIAL: NCT05677074
Title: Tolererer Fiske- og Skaldyrsallergikere Fiskeolietilskud? Et Klinisk Studie
Brief Title: Do Patients With Fish or Shellfish Allergy Tolerate the Consumption of Fish Oil Supplements? A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Lene Heise Garvey, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-22056640
Record Dates: First submitted 2022-12-20; First posted 2023-01-10 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Food Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity | interventions — Fish Oils; CVD protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolerance test of fish oil, cod oil, and krill oil (Experimental): All participants will have their tolerance of three different dietary supplements tested (fish oil, cod oil, and krill oil) using three methods: skin-prick-test, Basophil Histamine Release Assay, and oral provocation.
  Interventions: Dietary Supplement: Fish oil; Dietary Supplement: Cod oil; Dietary Supplement: Krill oil

INTERVENTIONS:
Dietary Supplement: Fish oil — The tolerance of fish oil is tested using three methods: skin-prick-test, Basophil Histamine Release Assay, and oral provocation.
Dietary Supplement: Cod oil — The tolerance of cod oil is tested using three methods: skin-prick-test, Basophil Histamine Release Assay, and oral provocation.
Dietary Supplement: Krill oil — The tolerance of krill oil is tested using two methods: skin-prick-test and Basophil Histamine Release Assay. (We were unable to acquire enough liquid krill oil to perform oral provocation with this supplement).

SUMMARY:
The purpose of this clinical study is to test whether patients with fish or shellfish allergy can ingest different types of fish oil supplements without having an allergic reaction.

To achieve this, the recruited participants will be asked to:

* provide a blood sample (used for Basophil Histamine Release Assay)
* undergo a skin-prick-test
* partake in multiple oral provocations

These three tests will indicate the likelihood that the participants can consume fish oil supplements without adverse allergic reactions (See the detailed description for an explanation of the tests).

The investigators will test the participants tolerance for three different types fish oil supplements: Fish oil, Cod liver oil, and krill oil.

DETAILED DESCRIPTION:
The Basophil Histamine Release Assay is a test that indicates whether or not the immune cells of the participant reacts when it comes into contact with the fish oils.

The skin-prick-test involves the participants having their skin exposed to the fish oils. This is done by first exposing a tiny needle to the given fish oil, and then pricking the needle into the skin on the forearm of the participant. In this way, the immune cells of the skin is exposed to the fish oils. If an allergic reaction occurs, the pricked skin will swell and turn reddish.

During the oral provocation, the participant is asked to ingest small, but increasing, doses of the fish oils over a period of 2 hours. The provocation will end when either an allergic reaction occurs or the participant has ingested a total dose of 5 mL fish oil.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Legally competent
* Understands Danish

Exclusion Criteria:

* Current use of antihistamine, immunosuppressants, and/or anti-IgE-treatment that cannot be safely terminated during the study period
* The presence of severe diseases such as: Cardiovascular disease, asthma, cancer, liver disease, kidney disease, hematological diseases, neurological diseases, dementia, immunological diseases, and endocrine diseases
* Chronic urticaria
* Severe atopic eczema
* Pregnancy and/or breastfeeding
* Participation in another clinical study the previous three months
* Known excessive use of alcohol and/or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Allergic reactions during fish oil provocation. | At 2 hours after the provocation or at the end of the provocation if terminated early (in case of allergic reaction).
  Presence of objective allergic symptoms (i.e. hives, redness, respiratory difficulties, and changes in blood pressure) during and two hours after the oral provocation.
Allergic reactions during cod oil provocation. | At 2 hours after the provocation or at the end of the provocation if terminated early (in case of allergic reaction).
  Presence of objective allergic symptoms (i.e. hives, redness, respiratory difficulties, and changes in blood pressure) during and two hours after the oral provocation.
Allergic reactions during krill oil provocation. | At 2 hours after the provocation or at the end of the provocation if terminated early (in case of allergic reaction).
  Presence of objective allergic symptoms (i.e. hives, redness, respiratory difficulties, and changes in blood pressure) during and two hours after the oral provocation.

SECONDARY OUTCOMES:
Skin-prick-test | 15 minutes after the skin-prick-test has been administered.
  The size of the hives are measured, if the diameter is >3 mm it is considered a positive result, if the negative and positive control are negative and positive, respectively
Basophil Histamine Release Assay | At baseline
  The histamine release when in contact with the fish oil is compared with the histamine release when in contact with the positive control: Phorbol 12-myristate 13-acetate (PMA) + ionomycin. A histamine release of >10% compared to the positive control is considered a positive result.
Subjective allergic symptoms during oral provocations | At 2 hours after each provocation or at the end of the provocation if terminated early (in case of allergic reaction).
  Subjective allergic symptoms (e.g. itchiness, throat irritation) are noted
Blood pressure during oral provocations | Change in blood pressure from baseline in case of allergic reaction
  Blood pressure (mmHg) is measured to detect possible changes from baseline,indicating the severity of an allergic reaction
Pulse during oral provocations | Change in blood pressure from baseline in case of allergic reaction
  Pulse (beats pr. min) is measured to detect possible changes from baseline, indicating the severity of an allergic reaction
Peak flow during oral provocations | Change in blood pressure from baseline in case of allergic reaction
  Peak flow (liters pr. minute) is measured to detect possible changes from baseline, indicating the severity of an allergic reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Gentofte Hospital, Gentofte Municipality, Hellerup, Denmark